CLINICAL TRIAL: NCT01378546
Title: Treatment of Lambert-Eaton Myasthenic Syndrome and Congenital Myasthenic Syndromes With 3, 4-Diaminopyridine
Brief Title: Treatment of Lambert-Eaton Myasthenic Syndrome (LEMS) With 3, 4 DAP
Status: No longer available | Type: Expanded Access
Sponsor: Louis H. Weimer, MD (Other)
Responsible Party: Sponsor-Investigator, Louis H. Weimer, MD, Clinical Professor of Neurology, Columbia University
Organization: Columbia University (Other)
Other Study IDs: AAAB2528
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Lambert Eaton Myasthenic Syndrome (LEMS)
MeSH Terms: conditions — Lambert-Eaton Myasthenic Syndrome | interventions — Amifampridine

INTERVENTIONS:
Drug: 3,4-diaminopyridine — Treatment will begin with 5mg three times a day or less.

SUMMARY:
Lambert Eaton Myasthenic Syndrome (LEMS) is rare neurological disorder that results in muscle weakness and limited reflex activity. More than half of LEMS cases are associated with a malignancy, usually small cell lung cancer, and tend to progress more quickly than cases not coupled with malignant cells.

3,4diaminopyridine (3,4DAP)is a drug that has been demonstrated to be effective in treating the weakness associated with LEMS as it increases strength and improves autonomic symptoms in LEMS patients. It is not currently approved by the FDA for use in the United States. The investigators plan to use 3,4DAP to treat patients with LEMS here at the Columbia University MDA/ALS Research Center.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with LEMS or a type of CMS likely to respond to 3, 4-DAP.
* If female of childbearing age, have negative pregnancy test, and be willing to practice and effective form of birth control during the study.
* Tested and found by ECG not to have a prolonged QTc syndrome.
* Agrees to have a second ECG at the time of peak drug effect. Has understood and signed the Informed Consent.

Exclusion Criteria:

* Is known to have a sensitivity to 3, 4-DAP.
* Has a history of past or current seizures or of severe asthma, or has an epileptiform EEG.
* Is believed by the investigator to be unable to comply with the protocol.
* Is unable to give informed consent.
* No patient will be excluded based on race, ethnicity, gender, or HIV status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-05; Primary Completion 2015-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Louis H Weimer, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States